CLINICAL TRIAL: NCT00393276
Title: Optimizing Vaccine Responsiveness in HIV-1 and HCV Infections by Identifying Determinants of Responsiveness: A Pilot Study
Brief Title: Determining Responses to Two Different Vaccines in HIV and HCV Infected Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A5232; 10154 (Registry Identifier: DAIDS ES Registry Number); 1R21AI066957-01 (NIH); ACTG A5232
Record Dates: First submitted 2006-10-25; First posted 2006-10-27 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hepatitis C
Keywords: Treatment Experienced; Treatment Naive; Immunizations
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — twinrix; Diphtheria-Tetanus Vaccine

ARMS (3):
- A (Experimental): HCV-infected defined as a positive result using polymerase chain reaction (PCR) without previous HCV-based therapy and without the presence of Child's B or C cirrhosis. These participants will be HIV-uninfected.
  Interventions: Biological: Twinrix; Biological: Decavac
- B (Experimental): HIV-infected and ARV naive, with a CD4 cell count of 300 cells/mm3 or greater, with no prior or current opportunistic infection, and with no indication for HIV therapy. These participants will be HCV-uninfected.
  Interventions: Biological: Twinrix; Biological: Decavac
- C (Experimental): HCV/HIV-coinfected as defined above in Arms A and B.
  Interventions: Biological: Twinrix; Biological: Decavac

INTERVENTIONS:
Biological: Twinrix — Combined hepatitis A and hepatitis B immunization
Biological: Decavac — Diphtheria and tetanus toxoid vaccine

SUMMARY:
Infection with either HIV or hepatitis C virus (HCV) affects immune system responses. The purpose of this study is to investigate the immune responses to two different vaccine formulations in HIV-infected, HCV-infected, and HCV/HIV- coinfected individuals.

DETAILED DESCRIPTION:
Individuals with HCV and HIV coinfection are especially hard to treat, and as a result, account for a high rate of deaths each year. Because HCV and HIV share transmission routes, HCV/HIV coinfection is common. Liver disease has emerged as a significant cause of death in individuals coinfected with HCV and HIV. Currently, the mechanisms by which HCV and HIV interact in HCV/HIV-coinfected individuals, including how these infections affect immune responses, are poorly understood. Research suggests that vaccination may prevent other comorbidities associated with HCV/HIV coinfection; however, responses to new vaccine antigens have been shown to be impaired in HCV or HIV-infected individuals. The purpose of this study is to identify the innate and adaptive immune defects present in HCV-infected, HIV-infected, and HCV/HIV-coinfected individuals. This study will evaluate whether these innate and adaptive immune defects predict responses to HBV neoantigen in the form of both a diphtheria/tetanus toxoid immunization (Decavac)and a hepatitis A-hepatitis B immunization (Twinrix).

This study will last approximately 24 weeks. Participants will be stratified to one of three arms, based on their HCV and HIV status:

* Arm A will enroll HCV-infected individuals who are HIV-uninfected
* Arm B will enroll HIV-infected individuals who are HCV-uninfected
* Arm C will enroll HCV/HIV-coinfected individuals

Arms B and C will open for enrollment before Arm A. Opening of enrollment for Arm A will be determined by the accrual progress of Arms B and C as evaluated by the ACTG Scientific Agenda Steering committee.

All participants will receive Decavac vaccination on Day 0, and a Twinrix vaccination on Days 0, 7, and 21. Study visits will occur around Days 0, 7, and 21, and at Weeks 6, 8, 12, and 24; all visits will include medical and medication history, blood collection, and a physical exam. Medication to treat HCV or HIV will not be provided by the study.

ELIGIBILITY:
Inclusion Criteria for Arm A Participants:

* HCV-infected
* HIV-uninfected

Inclusion Criteria for Arm B Participants:

* HIV-infected
* HCV-uninfected
* CD4 count greater than or equal to 300 cells/mm3 within 60 days prior to study entry

Inclusion Criteria for Arm C Participants:

* HIV-infected
* HCV-infected

Inclusion Criteria for All Participants:

* Documented hepatitis B virus (HBV) antibody status. If anti-HBV core antibody positive, documented HBV negative test within 30 days prior to study entry is required.
* Willing to use acceptable forms of contraception for the duration of the study and for 24 weeks after the last vaccination

Exclusion Criteria for Arm A Participants:

* Concurrent or recent treatment for HCV infection (within the past three months)

Exclusion Criteria for Arm B Participants:

* Current, prior, or clinical need for antiretroviral therapy (within the past three months prior to study entry)
* Opportunistic infection other than HCV

Exclusion Criteria for Arm C Participants:

* Concurrent or recent treatment for HCV infection (within the past three months)
* Current, prior, or clinical need for antiretroviral therapy (within the past three months prior to study entry). More information on this criterion can be found in the protocol.
* Opportunistic infection other than HCV

Exclusion Criteria for All Participants:

* History of exposure to hepatitis A vaccine, hepatitis B vaccine, or combined hepatitis A-hepatitis B vaccines
* Immunomodulatory agents for 7 days or more within 30 days prior to study entry. More information on this criterion can be found in the protocol.
* Concurrent immunizations (e.g., influenza, pneumococcal, other vaccine)within 3 days prior to study entry
* Active or recent (in the last six months prior to study entry) CDC Category C event. More information on this criterion can be found in the protocol
* Systemic anticancer chemotherapy or radiation within 24 weeks prior to study entry, or anticipated need to begin such treatment
* Past or current immunologically-mediated disease. More information on this criterion can be found in the protocol.
* Current bacterial infection requiring treatment, therapy, or hospitalization within 1 week prior to study entry
* Serious illness requiring systemic treatment and/or hospitalization. Participants who complete therapy or are clinically stable on therapy for at least 14 days prior to study entry are not excluded.
* Current uncontrolled seizure disorders
* Active bleeding varices, or Child's B or C cirrhosis. More information on this criterion can be found in the protocol.
* Serious bleeding disorder that poses a risk to a participant for intramuscular injections
* Known allergy or sensitivity to study vaccines or their formulations
* Current drug or alcohol use that, in the opinion of the investigator, interferes with study participation
* Pregnant or breastfeeding
* Use of systemic investigational agents within 30 days prior to entry
* History of any hepatitis A vaccine within one year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
B-cell humoral responses | At Week 8
T-cell responses as reflected by hepatitis B and tetanus antibody titers | At Week 8
Dendritic cell, B-cell, and T-cell functional markers | At Study Entry

SECONDARY OUTCOMES:
B-cell functional marker | At Week 6
T-cell responses to hepatitis A, hepatitis B, and tetanus antigens | At Weeks 3 and 8
Longitudinal serum antibody titers to hepatitis A, hepatitis B, and tetanus (B-cell responses) | At Study Entry and Weeks 1, 3, 6, 8, 12, and 24
CD4/CD8 and HCV genotype | At Study entry
Baseline antibody status for hepatitis B core antigen (anti-HBc) | At Study entry

CONTACTS AND LOCATIONS:
Overall Officials: Donald D. Anthony, MD, PhD, Study Chair — Case Western Reserve University; Benigno Rodriguez, MD, Study Chair — Division of Infectious Diseases, University Hospital of Cleveland
Locations (12):
- United States (11):
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Massachusetts General Hospital Clinical Research Site (MGH CRS) CRS, Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Trinity Health and Wellness Center CRS, Dallas, Texas
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Maier I, Wu GY. Hepatitis C and HIV co-infection: a review. World J Gastroenterol. 2002 Aug;8(4):577-9. doi: 10.3748/wjg.v8.i4.577. PMID 12174359
- [Background] Rockstroh JK. Management of hepatitis B and C in HIV co-infected patients. J Acquir Immune Defic Syndr. 2003 Sep;34 Suppl 1:S59-65. doi: 10.1097/00126334-200309011-00009. PMID 14562859
- [Background] Sulkowski MS, Mast EE, Seeff LB, Thomas DL. Hepatitis C virus infection as an opportunistic disease in persons infected with human immunodeficiency virus. Clin Infect Dis. 2000 Apr;30 Suppl 1:S77-84. doi: 10.1086/313842. PMID 10770916